CLINICAL TRIAL: NCT05635708
Title: Master Protocol: A Phase 2, Open-label, Multi-arm Study of Tislelizumab in Combination With Investigational Agents With or Without Chemotherapy in Patients With Previously Untreated, Locally Advanced, Unresectable, or Metastatic Non-Small Cell Lung Cancer
Brief Title: A Study of Tislelizumab in Combination With Investigational Agents in Participants With Non-Small Cell Lung Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: BeiGene (Industry)
Responsible Party: Sponsor
Organization: BeOne Medicines (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BGB-LC-201; CTR20230892 (Other: ChinaDrugTrials); 2022-502738-18-00 (EU CTIS Number)
Record Dates: First submitted 2022-11-23; First posted 2022-12-02 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Non-small Cell Lung Cancer; Metastatic Non-small Cell Lung Cancer
Keywords: Non-small Cell Lung Cancer; NSCLC; programmed cell death protein-1; PD-L1 Low Tumors; PD-L1 Negative Tumors; Metastatic Non-Small Cell Lung Cancer; PD-L1 High Tumors
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — tislelizumab; Carboplatin; Cisplatin; Pemetrexed; Paclitaxel; Taxes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- Sub-study 1: Arm 1A (Experimental): Tislelizumab + BGB-A445
  Interventions: Drug: Tislelizumab; Drug: BGB-A445
- Sub-study 1: Arm 2A (Experimental): Tislelizumab + LBL-007
  Interventions: Drug: Tislelizumab; Drug: LBL-007
- Sub-study 1: Arm 3A (Experimental): Tislelizumab + BGB-15025
  Interventions: Drug: Tislelizumab; Drug: BGB-15025
- Sub-study 1: Reference Arm Tislelizumab alone (Active Comparator): Tislelizumab alone
  Interventions: Drug: Tislelizumab
- Sub-study 2: Arm 1B (Experimental): Tislelizumab + investigator's choice of histology-appropriate chemotherapy + BGB-A445
  Interventions: Drug: Tislelizumab; Drug: BGB-A445; Drug: Carboplatin; Drug: Cisplatin; Drug: pemetrexed; Drug: Paclitaxel; Drug: Nab paclitaxel
- Sub-study 2: Arm 2B (Experimental): Tislelizumab + investigator's choice of histology-appropriate chemotherapy + LBL-007
  Interventions: Drug: Tislelizumab; Drug: LBL-007; Drug: Carboplatin; Drug: Cisplatin; Drug: pemetrexed; Drug: Paclitaxel; Drug: Nab paclitaxel
- Sub-study 2: Arm 3B (Experimental): Tislelizumab + investigator's choice of histology-appropriate chemotherapy + BGB-15025
  Interventions: Drug: Tislelizumab; Drug: Carboplatin; Drug: Cisplatin; Drug: pemetrexed; Drug: Paclitaxel; Drug: Nab paclitaxel; Drug: BGB-15025
- Sub-study 2: Reference Arm (Active Comparator): Tislelizumab + investigator's choice of histology-appropriate chemotherapy
  Interventions: Drug: Tislelizumab; Drug: Carboplatin; Drug: Cisplatin; Drug: pemetrexed; Drug: Paclitaxel; Drug: Nab paclitaxel

INTERVENTIONS:
Drug: Tislelizumab — Administered by intravenous infusion
Drug: BGB-A445 — Administered by intravenous infusion
  Arms: Sub-study 1: Arm 1A; Sub-study 2: Arm 1B
Drug: LBL-007 — Administered by intravenous infusion
  Arms: Sub-study 1: Arm 2A; Sub-study 2: Arm 2B
Drug: Carboplatin — Investigator's choice; administered by intravenous infusion
  Arms: Sub-study 2: Arm 1B; Sub-study 2: Arm 2B; Sub-study 2: Arm 3B; Sub-study 2: Reference Arm
Drug: Cisplatin — Investigator's choice; administered by intravenous infusion
  Arms: Sub-study 2: Arm 1B; Sub-study 2: Arm 2B; Sub-study 2: Arm 3B; Sub-study 2: Reference Arm
Drug: pemetrexed — Investigator's choice; administered by intravenous infusion
  Arms: Sub-study 2: Arm 1B; Sub-study 2: Arm 2B; Sub-study 2: Arm 3B; Sub-study 2: Reference Arm
Drug: Paclitaxel — Investigator's choice; administered by intravenous infusion
  Arms: Sub-study 2: Arm 1B; Sub-study 2: Arm 2B; Sub-study 2: Arm 3B; Sub-study 2: Reference Arm
Drug: Nab paclitaxel — Investigator's choice; administered by intravenous infusion
  Arms: Sub-study 2: Arm 1B; Sub-study 2: Arm 2B; Sub-study 2: Arm 3B; Sub-study 2: Reference Arm
Drug: BGB-15025 — Administered Orally
  Arms: Sub-study 1: Arm 3A; Sub-study 2: Arm 3B

SUMMARY:
The purpose of this study is to assess the antitumor activity, safety, and tolerability of tislelizumab plus investigational agent(s) with or without chemotherapy. This study is structured as a master protocol with separate sub- studies. Sub-study 1 includes participants with non-small cell lung cancer (NSCLC) with high programmed cell death protein ligand-1 (PD-L1) expression (≥ 50%), and Sub-study 2 includes participants with NSCLC with low or negative (PD-L1) expression (< 50%).

ELIGIBILITY:
Key Inclusion Criteria:

1. Histologically or cytologically confirmed non-small cell lung cancer (NSCLC), including nonsquamous or squamous subtypes, that is either locally advanced or recurrent and not eligible for curative surgery and/or definitive chemoradiotherapy, or metastatic NSCLC.
2. No prior systemic therapy administered as the primary treatment for metastatic NSCLC. Prior adjuvant or neoadjuvant chemotherapy, definitive chemoradiation, or adjuvant radiotherapy for locally advanced disease is permitted, provided the last dose of chemotherapy and/or radiotherapy occurred at least 6 months prior to randomization/enrollment.
3. Tumor programmed death-ligand 1 (PD-L1) expression must be evaluable, as determined by a local or central laboratory using archival tumor tissue or a fresh biopsy. Participants with unknown PD-L1 expression are not eligible.
4. At least one measurable lesion, as defined by Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1.
5. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1.

Key Exclusion Criteria:

1. Diagnosis of mixed small cell lung cancer.
2. Known genomic alterations for which effective targeted therapies are available according to local standard of care, including but not limited to:

   * Epidermal growth factor receptor (EGFR) mutations
   * Anaplastic lymphoma kinase (ALK) rearrangements
   * B-Raf proto-oncogene (BRAF) mutations
   * Rearranged during transfection (RET) fusions
   * c-ros oncogene 1 (ROS1) rearrangements
3. Participants with nonsquamous NSCLC and unknown EGFR mutation status must undergo local testing. Those found to have EGFR-sensitizing mutations will be excluded.
4. Prior treatment with immune-based therapies that target immune checkpoint pathways, including:

   * PD-1 (programmed cell death protein 1) inhibitors
   * PD-L1 (programmed death-ligand 1) inhibitors
   * PD-L2 (programmed death-ligand 2) inhibitors
   * TIGIT (T cell immunoreceptor with Ig and ITIM domains) inhibitors
   * LAG-3 (lymphocyte activation gene 3) inhibitors
5. Participants previously treated with these agents in a neoadjuvant, adjuvant, or consolidation setting may be eligible if a treatment-free interval of at least 6 months has elapsed since the last dose and radiologic evidence of recurrence is present.
6. Use of Chinese herbal medicines or Chinese patent medicines intended for cancer control within 14 days prior to randomization/enrollment.
7. Presence of active leptomeningeal disease, untreated or uncontrolled brain metastases, or active autoimmune disease.

Note: Additional protocol-defined and sub-study-specific criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2023-03-07 (Actual); Primary Completion 2025-12-31 (Actual); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Confirmed overall response rate (ORR) | Up to 6 months
  ORR is defined as the percentage of participants with partial or complete response, as assessed by the investigator using the Response Evaluation Criteria in Solid Tumors (RECIST) Version (v)1.1

SECONDARY OUTCOMES:
Progression-free survival (PFS) | Up to 1 year
  PFS is defined as the time from date of randomization, or the first dose for safety lead-in participants , until first documentation of progression or death, whichever comes first, as assessed by the investigator using RECIST v1.
Duration of Response (DOR) | Up to 1 year
  DOR is defined as the time from the first determination of a confirmed response per RECIST v1.1 until the first documentation of progression or death, whichever comes first as assessed by the investigator
Clinical Benefit Rate (CBR) | Up to 6 months
  CBR is defined as the percentage of participants with a best overall response of a complete response, partial response, or durable stable disease, as assessed by the investigator using RECIST v1.1
Disease Control Rate (DCR) | Up to 6 months
  DCR is defined as the percentage of participants with a best overall response of complete response, partial response, or stable disease, as assessed by the investigator using RECIST v1.1
Number of participants with adverse events (AEs) | From the first dose of study drug(s) to 90 days after initiation of new anticancer therapy, death, withdrawal of consent, or loss to follow-up, whichever occurs first, up to approximately 2 years
  Number of participants with treatment-emergent adverse events (TEAEs) and serious adverse events (SAEs), including laboratory values, vital signs, physical examination findings, and electrocardiogram results.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — BeiGene
Locations (61):
- United States (5):
  - Valkyrie Clinical Trials, Los Angeles, California
  - Massachusetts General Hospital, Boston, Massachusetts
  - Memorial Sloan Kettering Cancer Center Mskcc, New York, New York
  - Providence Portland Medical Center, Portland, Oregon
  - The University of Texas Md Anderson Cancer Center, Houston, Texas
- Australia (6):
  - Blacktown Cancer and Haematology Centre, Blacktown, New South Wales
  - Chris Obrien Lifehouse, Camperdown, New South Wales
  - Northern Beaches Hospital, Frenchs Forest, New South Wales
  - Port Macquarie Base Hospital, Port Macquarie, New South Wales
  - One Clinical Research, Nedlands, Western Australia
  - St John of God Health Care, Subiaco, Western Australia
- Brazil (5):
  - Hospital de Amor Barretos, Barretos
  - Hospital Do Cancer de Londrina, Londrina
  - Centro Gaucho Integrado de Oncologia Hospital Mae de Deus, Porto Alegre
  - Fundacao Faculdade Regional de Medicina de Sao Jose Do Rio Preto, São José do Rio Preto
  - Icesp Instituto Do Cancer Do Estado de Sao Paulo Octavio Frias de Oliveira, São Paulo
- Cross Cancer Institute, Edmonton, Alberta, Canada
- China (18):
  - The Second Hospital of Anhui Medical University, Hefei, Anhui
  - The Fifth Medical Center of Chinese Pla General Hospital, Beijing, Beijing Municipality
  - Fujian Cancer Hospital, Fuzhou, Fujian
  - Affiliated Hospital of Hebei University, Baoding, Hebei
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Hubei Cancer Hospital, Wuhan, Hubei
  - Nantong Tumor Hospital Branch North, Nantong, Jiangsu
  - The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - The First Affiliated Hospital of Nanchang University Branch Xianghu, Nanchang, Jiangxi
  - Jining No Peoples Hospital East Branch, Jining, Shandong
  - Linyi Peoples Hospital, Linyi, Shandong
  - Affiliated Zhongshan Hospital of Fudan University, Shanghai, Shanghai Municipality
  - Shanghai East Hospital Branch Hospital, Shanghai, Shanghai Municipality
  - Shanghai Pulmonary Hospital, Shanghai, Shanghai Municipality
  - Shanxi Provincial Cancer Hospital, Taiyuan, Shanxi
  - Tianjin Medical University Cancer Institute and Hospital, Tianjin, Tianjin Municipality
  - Taizhou Hospital of Zhejiang, Taizhou, Zhejiang
- France (2):
  - Institut Curie, Paris
  - Chu Nantes Hopital Nord Laennec, SaintHerblain
- Arensia Exploratory Medicine Llc, Tbilisi, Georgia
- Italy (2):
  - Regina Elena, Istituto Nazionale Dei Tumori, Ifo, Irccs, Roma
  - Centro Ricerche Cliniche Di Verona, Verona
- Malaysia (3):
  - Pulau Pinang Hospital, George Town
  - Tengku Ampuan Afzan Hospital, Kuantan
  - Sarawak General Hospital, Kuching
- The Institute of Oncology, Arensia Exploratory Medicine, Chisinau, Moldova
- Romania (2):
  - Institute of Oncology Bucharest Prof Dr Alexandru Trestioreanu, Bucureti
  - Arensia Research Clinic At the Oncology Institute Prof Dr Ion Chiricu, ClujNapoca
- National Cancer Centre Singapore, Singapore, Singapore
- South Korea (7):
  - Chungbuk National University Hospital, Cheongju-si, Chungcheongbukdo
  - Seoul National University Bundang Hospital, BundangGu SeongnamSi, Gyeonggi-do
  - National Cancer Center (Korea), IlsandongGu GoyangSi, Gyeonggi-do
  - The Catholic University of Korea, St Vincents Hospital, PaldalGu SuwonSi, Gyeonggi-do
  - Samsung Medical Center, GangnamGu, Seoul Teugbyeolsi
  - Severance Hospital Yonsei University Health System, SeodaemunGu, Seoul Teugbyeolsi
  - Asan Medical Center, SongpaGu, Seoul Teugbyeolsi
- Spain (3):
  - Hospital Universitario Vall Dhebron, Barcelona
  - Hospital Universitario de Octubre, Madrid
  - Hospital Universitario Virgen Del Rocio, Seville
- Thailand (4):
  - Songklanagarind Hospital (Prince of Songkhla University), Hat Yai
  - Srinagarind Hospital (Khon Kaen University), Muang
  - Maharaj Nakorn Chiang Mai Hospital (Chiang Mai University), Muang
  - Hrh Princess Maha Chakri Sirindhorn Medical Center (Srinakharinwirot University), Ongkharak

IPD SHARING:
Plan to Share IPD: Yes
BeiGene shares data on completed studies responsibly and provides qualified scientific and medical researchers access to data and supporting documentation for clinical trials in dossiers for medicines and indications after submission and approval in the United States, China, and Europe. Clinical trials supporting subsequent local approvals, new indications, or combination products are eligible for sharing once corresponding regulatory approvals are achieved.
  BeiGene shares data only when permitted by applicable data privacy and security laws and regulations, when it is feasible to do so without compromising the privacy of study participants, and other considerations.
  Qualified researchers with appropriate competencies who are engaged in novel scientific research may submit a request for participant-level data with a research proposal for BeiGene review. Research teams must include a biostatistician and sign a Data Sharing Agreement prior to receiving access to clinical trial data.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: See plan description
Access Criteria: See plan description
URL: https://beigene.com/science/clinical-trials/